CLINICAL TRIAL: NCT00875186
Title: Impact of Aerobic Physical Exercising on Body Composition and co-Morbidities in Patients After Laparoscopic Roux-en-Y Gastric Bypass
Brief Title: The Influence of Aerobic Endurance Training After Roux-en-Y-Gastric Bypass
Acronym: AET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Assoc. Professor Edward Shang, MD, Department of Surgery, University Hospital Mannheim
Other Study IDs: AET 1
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Morbid Obesity
Keywords: bariatric surgery; co-morbidities; aerobic physical exercise
MeSH Terms: conditions — Obesity, Morbid | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- multiple-exercise group (ME): participants exercised 2 times weekly for 1 hour (aerobic endurance training)
  Interventions: Other: aerobic endurance training
- Low-exercise group (LE): participants exercises 1 time weekly for 1 hour (aerobic endurance training)
  Interventions: Other: aerobic endurance training

INTERVENTIONS:
Other: aerobic endurance training — participants exercises 2 times weekly for 1 hour (aerobic endurance training)
  Other Names: aerobic physical exercise
  Groups: multiple-exercise group (ME)
Other: aerobic endurance training — participants exercised 1 time weekly for 1 hour (aerobic endurance training)
  Other Names: aerobic physical exercise
  Groups: Low-exercise group (LE)

SUMMARY:
The aim of this study was to assess the efficiency of aerobic physical exercise (APE) on weight loss, body composition and co-morbidities in patients after laparoscopic Roux-en-Y Gastric bypass (RYGBP).

DETAILED DESCRIPTION:
The only effective treatment for patients with morbid obesity is bariatric surgery. Sudden weight loss following bariatric operations for morbid obesity, such as Roux-en-Y gastric bypass (RYGBP) can result in a concurrent decrease in lean body mass. However the long-time results (weight reduction, elimination co-morbidities) are depending on the post operative treatment. Aerobic physical exercising (APE) is well accepted in conservative treatment of obesity as well as of diabetes mellitus type 2 (DM). The aim of this study was to assess the efficiency of APE on weight loss, body composition and co-morbidities in patients after laparoscopic Roux-en-Y Gastric bypass (RYGBP).

ELIGIBILITY:
Inclusion Criteria:

* Obesity WHO III

Exclusion Criteria:

* Contraindications of aerobic endurance training

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: morbidly obese patients underwent laparoscopic Roux-en-Y gastric bypass as a primary procedure for morbid obesity
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2006-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
effects of aerobic physical exercising (APE) on weight loss | 10 years

SECONDARY OUTCOMES:
effects of aerobic physical exercising (APE) on co-morbidities | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Edward Shang, M.D., Study Chair — Universitätsmedizin Mannheim; Till Hasenberg, M.D., Principal Investigator — Universitätsmedizin Mannheim
Locations (1):
- Department of Surgery, University Hospital Mannheim, Mannheim, Germany